CLINICAL TRIAL: NCT06371313
Title: Endocrine, Metabolic and Inflammatory Characteristics of Offspring of Mothers With PCOS Hyperandrogenism: A Cross-sectional Study
Brief Title: Endocrine, Metabolic and Inflammatory Characteristics of Offspring of Mothers With PCOS Hyperandrogenism
Status: Completed | Type: Observational
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Li Li, Deputy Director, Institute of Women's and Children's Health, Guangdong Women and Children Hospital
Other Study IDs: GuangdongWCH-LiLi03
Record Dates: First submitted 2024-04-07; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: PCOS
Keywords: PCOS; Hyperandrogenemia; Offspring; Endocrine and Metabolism; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cord Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HA Group: Maternal hyperandrogenism of PCOS women with full-term singleton delivery were selected, and umbilical cord blood of their newborns was collected.
- Control Group: Healthy pregnant women with full-term singleton delivery were randomly selected, and umbilical cord blood of their newborns was collected.

SUMMARY:
This study is a cross-sectional study to explore the endocrine metabolism and inflammatory characteristics of the offspring of mothers with PCOS hyperandrogenism, in order to provide a theoretical basis for finding the cause of PCOS.

DETAILED DESCRIPTION:
This study randomly selected 20 women with PCOS and hyperandrogenism who gave birth to a singleton at term at Guangdong Maternal and Child Health Hospital from May 2023 to March 2024, and set them as the HA group. In addition, 22 healthy women were randomly selected as controls. group, the fasting blood glucose (FPG) level of the newborn's peripheral blood and the androgen, fasting insulin and inflammatory factor levels of the newborn's umbilical cord blood were collected respectively.

Among them, the detection indicators of newborn umbilical cord blood include testosterone (T), androstenedione (AND), dehydroepiandrosterone sulfate (DHEA-S), sex hormone binding globulin (SHBG), free androgen index (FAI), Fasting insulin (FINS), white blood cell count (WBC), neutrophil count (NEUT), high-sensitivity C-reactive protein (hs-CRP), and interleukin (IL)-6.

All collected data were statistically analyzed to compare the differences in levels of androgens, fasting insulin, and inflammatory factors in the umbilical cord blood of newborns in the HA group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of polycystic ovary syndrome patients must meet the Rotterdam criteria.
* Aged between 18 and 45 years old.
* The gestational age of delivery is between 37 and 41 weeks of gestation.
* Hyperandrogenemia inclusion criteria: elevated peripheral blood androgens, including testosterone, androstenedione, and dehydroepiandrosterone sulfate.
* Singleton pregnancy.
* Signed informed consent form.

Exclusion Criteria:

* Combined with reproductive organ malformations or chromosomal abnormalities.
* Combined with chronic diseases such as diabetes and hypertension.
* Combined with thyroid disease or other serious systemic diseases such as cardiovascular disease.
* Multiple pregnancy.
* Combined with congenital adrenal hyperplasia, Cushing's syndrome, hypertension Prolactinoma, and androgen-secreting tumor-related diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The women selected into the study group were diagnosed with PCOS before pregnancy and were complicated with hyperandrogenism.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Testosterone | Within one year after neonatal cord blood collection.
  Testosterone is one of the androgens, which can be used to assess androgen levels.
Androstenedione | Within one year after neonatal cord blood collection.
  Androstenedione is one of the androgens, which can be used to assess androgen levels.
Dehydroepiandrosterone Sulfate | Within one year after neonatal cord blood collection.
  Dehydroepiandrosterone Sulfate is one of the androgens, which can be used to assess androgen levels.
Sex Hormone Hinding Globulin | Within one year after neonatal cord blood collection.
  Sex hormone-binding globulin, also known as testosterone-estradiol binding globulin, is a carrier of sex hormones and can reflect the level of sex hormones.
Free Androgen Index | Within one year after neonatal cord blood collection.
  The free androgen index can reflect the biological activity of androgen.
Fasting Insulin | Within one year after neonatal cord blood collection.
  Insulin is a hormone secreted by pancreatic beta cells that lowers blood glucose and produces energy metabolism. Its level can assist in the diagnosis of insulin resistance.
White Blood Cell Count | Within six hours of neonatal cord blood collection.
  The white blood cell count can assess the inflammatory status.
Neutrophil Count | Within six hours of neonatal cord blood collection.
  Neutrophil count can be used to assess the inflammatory status.
High-sensitivity C-reactive Protein | Within six hours of neonatal cord blood collection.
  High-sensitivity C-reactive protein can be used to assess the inflammatory status.
Interleukin-6 | Within one year after neonatal cord blood collection.
  Interleukin (IL)-6 can be used to assess the inflammatory status.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, M.D., Study Chair — Guangdong Women and Children Hospital; Chen Yuan, Master, Principal Investigator — Guangdong Women and Children Hosptial
Locations (1):
- Guangdong Women and Children Hosptial, Guanzhou, Guangdong, China